CLINICAL TRIAL: NCT04261179
Title: An Exploratory Prospective, Open-label, Unicentric Study With Cross-over Design, Comparing Lymphoseek® vs. Albumin Nanocolloid for Image- Guided Sentinel Lymph Node Mapping in Head and Neck, Melanoma and Breast Cancer.
Brief Title: Study Comparing Lymphoseek® vs. Albumin Nanocolloid in Head and Neck, Melanoma and Breast Cancer
Acronym: SENTINELSEEK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Project Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-003825-56
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Head Cancer; Neck Cancer; Melanoma; Breast Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Melanoma; Breast Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran; technetium Tc 99m nanocolloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphoseek + Nanocoll (Other): Comparison of the concordance of albumin nanocolloid and Lymphoseek® in the detection of lymph nodes of primary and secondary stage drainage by performing two lymphogammagrams
  Interventions: Drug: Lymphoseek; Drug: Nanocoll

INTERVENTIONS:
Drug: Lymphoseek — 50 μg microgram(s), timepoint: 30-60 minutes
Drug: Nanocoll — 500 μg microgram(s), timepoint: 30-60 minutes

SUMMARY:
Comparison of the concordance of albumin nanocolloid and Lymphoseek® in the detection of lymph nodes of primary and secondary stage drainage by performing two lymphogammagrams

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed diagnosis of melanoma, breast cancer or head and neck cancer and candidate for surgical resection with lymph node mapping being a part of the surgical plan.
* At least 18 years of age at the time of consent.
* The subject is clinically node negative (cN0) at the time of screening.
* In Melanoma Patients

  * Diagnosis of primary melanoma with sentinel node indication ( >0.8 mm Breslow thickness; clinically negative lymph nodes)
* In Breast Cancer Patients

  * T1-T2 N0 breast cancer.
  * Patients with pure ductal carcinoma in situ (DCIS) if lymph node biopsy is part of the surgical plan.
* In Oral cavity tumors patients

  * T1-T2 N0 oral cavity squamous cell carcinoma

Exclusion Criteria:

* Pregnancy or lactation
* Clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes
* Patients that have had preoperative chemotherapy, immunotherapy or radiation therapy
* Patients who have undergone node basin surgery of any type or radiation to the nodal basin(s) potentially draining the primary tumor
* Patients who have undergone a wide excision for their tumor or complex reconstruction (rotation, free flap or skin graft of any type).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Nodal Concordance: proportion of lymph nodes identified by 99mTc-tilmanocept vs nanocolloidal human serum albumin by lymphoscintigraphies | for at least 48 consecutive hours
  number and diameter in millimeters of nodes affected identified by 99mTc-tilmanocept vs nanocolloidal

SECONDARY OUTCOMES:
Time frame to ascertain the sentinel nodes | 1 week
Concordance among early and delayed images obtained withLymphoseek® or with albumianocolloid and the SPECT/CT images. | 1 week
Number of sentinel nodes and secondary nodes depicted | 1 week
Tracer retention in injection site | 1 week
Safety and tolerability of 99mTctilmanocept (Lymphoseek®) | 1 week
  Number of participants with treatment-related adverse events as assessed by Lymphoseek® or with albuminanocolloid

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico y provincial de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No